CLINICAL TRIAL: NCT06383130
Title: A Pragmatic Diagnostic Accuracy Study of a Triple Diagnostic Approach and Exploratory Biomarkers in Adult Asthma Diagnosis
Brief Title: London Asthma Diagnostics Study
Acronym: LADS
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Asthma UK (Other); General Practitioners Research Institute (Network)
Responsible Party: Sponsor
Other Study IDs: 24SM8792
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oscillometry with reversibility testing — Oscillometry is a test that uses sound waves to measure the mechanical properties in the lungs during tidal breathing
Diagnostic Test: Breath volatile testing — We will be optimising and evaluating the sensitivity and specificity of a novel breath volatile organic compound test of a combination of reactive aldehydes using a gas chromatography-ion mobility spectrometry device
Diagnostic Test: Nasal eosinophil peroxidase — We will be evaluating the sensitivity and specificity of a novel nasal swab test for eosinophil peroxidase
Diagnostic Test: Handheld capnometry — We will be evaluating handheld capnometry (carbon dioxide breath testing) to diagnose adult asthma

SUMMARY:
The goal of this trial is to learn if the addition of oscillometry with reversibility testing increases diagnostic accuracy in adult asthma diagnosis, when added to current standard of care tests: spirometry with reversibility testing and Fractional Exhaled Nitric Oxide (FeNO). The main question it aims to answer is:

- Does oscillometry with reversibility testing increase diagnostic accuracy in detection of asthma in adults when added to spirometry with reversibility and FeNO?

Researchers will evaluate the diagnostic accuracy of this approach with the reference standard, which is a clinically adjudicated diagnosis of asthma by two respiratory clinicians based on history and investigation results.

Participants will

* Undergo oscillometry testing alongside their routine asthma investigations within their scheduled clinic visit
* Optionally participate in our sub-studies on new breath and nasal swab tests for asthma
* Optionally participate in our qualitative substudy on patients views and attitudes to asthma testing and oscillometry

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by GP with either (a) possible incident asthma or (b) a diagnostic label of asthma without prior confirmatory objective diagnosis
* Age≥18 years
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study
* Able to give informed consent

Exclusion Criteria:

* Age <18 years
* A chest infection or exacerbation requiring antibiotics or steroids within 4 weeks of testing
* Contraindications to spirometry testing
* Established or coded diagnosis of COPD
* Pregnancy or lactating
* Other medical condition that in the opinion of the investigator would preclude compliance with the study protocoll
* Inability to understand English
* Involvement in Clinical Trial of an Investigational Medicinal Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be eligible if being referred by their doctor for investigation for possible asthma, or for confirmation of asthma due to absence of objective diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy (sensitivity, specificity) of a combination of oscillometry ± reversibility, spirometry ± reversibility and FeNO | 6 months
  To evaluate the diagnostic accuracy (sensitivity, specificity) of a combination of oscillometry ± reversibility, spirometry ± reversibility and FeNO for adult asthma diagnosis compared to the diagnostic reference standard.

SECONDARY OUTCOMES:
To conduct an analysis comparing the diagnostic accuracy of (i) oscillometry ± reversibility with spirometry ± reversibility, (ii) spirometry±reversibility with FeNO and (iii) oscillometry ±reversibility and FeNO | 6 months
  To compare the sensitivity and specificity of pairwise permutations of testing
To compare the concordance of positive and negative test results for (i) oscillometry±reversibility, (ii) spirometry ±reversibility and (iii) Fractional Exhaled Nitric Oxide (FeNO) | 6 months
  To assess the degree of agreement between each of the diagnostic tests
To collect data on (i) testing time, (ii) testing burden, (iii) general feasibility of implementation of the asthma diagnostic tests | 6 months
  We will collect data on feasibility on each of the diagnostics (spirometry, FeNO, oscillometry)

OTHER OUTCOMES:
To evaluate the diagnostic accuracy of the targeted reactive aldehyde species (RASP) panel in breath for asthma diagnosis | 6 months
  As an exploratory endpoint we will be optimising and assessing the diagnostic accuracy of a novel breath volatile organic compound test in asthma
To evaluate the diagnostic accuracy of nasal biomarker eosinophil peroxidase (EPX) | 6 months
  As an exploratory endpoint we will be assessing the diagnostic accuracy of a novel nasal swab eosinophil protein biomarker for asthma
To evaluate the diagnostic accuracy of tidal breath CO2 waveforms using the N-Tidal handheld capnometry device | 6 months
  As an exploratory endpoint we will be assessing the diagnostic accuracy of handheld capnometry for asthma

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No